CLINICAL TRIAL: NCT00617123
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Ocular Safety of SCH 530348 in Subjects Participating in the Schering-Plough P04737 Study (TRA^SM-Secondary Prevention Ocular Safety Study)
Brief Title: Trial to Assess the Ocular Safety of Vorapaxar (SCH 530348) in Participants With Atherosclerosis (Study P05183)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: The TIMI Study Group (Other); Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: P05183; MK-5348-018 (Other: Merck Protocol Number)
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Results first posted 2014-07-14 (Estimated); Last update posted 2018-09-21 (Actual); Status verified 2018-08

CONDITIONS: Atherosclerosis; Ischemia; Myocardial Infarction; Cerebrovascular Accident
MeSH Terms: conditions — Atherosclerosis; Ischemia; Myocardial Infarction; Stroke | interventions — vorapaxar

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vorapaxar (Experimental): Participants receive a vorapaxar 2.5 mg tablet administered orally once daily for 1 year
  Interventions: Drug: Vorapaxar 2.5 mg
- Placebo (Placebo Comparator): Participants receive a matching placebo tablet to vorapaxar administered orally once daily for 1 year
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vorapaxar 2.5 mg — Vorapaxar 2.5 mg oral tablet
  Arms: Vorapaxar
Drug: Placebo — matching placebo oral tablet
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the long-term ocular safety of SCH 530348 (vorapaxar) in participants with established atherosclerotic disease who are enrolled into the TRA 2°P - TIMI 50 Study (P04737) (NCT00526474).

ELIGIBILITY:
Inclusion Criteria:

* Evidence or a history of atherosclerosis involving the coronary, cerebral, or peripheral vascular systems

Exclusion Criteria:

* The study will include participants who meet none of the exclusion criteria for the parent protocol (P04737) and also the following:

  * history or evidence of age-related macular degeneration on baseline evaluation
  * history of diabetic macular edema, or evidence of treated diabetic retinopathy on baseline evaluation
  * history or evidence of other retinal diseases, including retinal injury, on baseline evaluation
  * history or evidence of retinal surgery, including laser photocoagulation, on baseline evaluation
  * history or evidence of glaucoma on baseline evaluation
  * history or evidence of high intraocular pressure of >22 mm Hg on baseline evaluation
  * evidence of center foveal thickness of >190 µm on baseline OCT examination
  * presence of vacuoles in the retina on baseline OCT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2008-07-01 (Actual); Primary Completion 2010-10-01 (Actual); Study Completion 2010-10-01 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=P05183&kw=P05183&tab=access

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from participants enrolled in Study SCH 530348 P04737 (NCT00526474) and met the inclusion/exclusion criteria for this study.
Pre-assignment Details: A total of 258 particpants were referred to opthalmology sites, 65 of whom did not particpate in this study (P05138) beyond the screening visit and were not included in the analysis of ocular safety. A total of 193 participants were included in the analysis of ocular safety.
Period: Referral Screening Period
Arm/Group | Vorapaxar | Placebo
Started | 137 | 121
Completed | 98 | 95
Not Completed | 39 | 26
Not completed — Did Not Meet Protocol Eligibility | 36 | 24
Not completed — Did Not Wish To Continue | 3 | 1
Not completed — Adverse Event | 0 | 1
Period: Study Treatment Period
Arm/Group | Vorapaxar | Placebo
Started | 98 | 95
Treated | 97 (1 participant was not treated) | 95
Completed | 81 | 79
Not Completed | 17 | 16
Not completed — Withdrawal by Subject | 8 | 12
Not completed — Adverse Event | 7 | 3
Not completed — Did Not Meet Protocol Eligibility | 2 | 0
Not completed — Noncompliance with Protocol | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants who were included in the analysis of ocular safety.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vorapaxar | Placebo | Total
Number analyzed (Participants) | 98 | 95 | 193
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (10.1) | 55.3 (11.7) | 55.9 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 26 | 53
  Male | 71 | 69 | 140

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Develop Vacuolization in the Inner Nuclear Layer (INL) of the Retina as Measured by Ocular Coherence Tomography (OCT)
Description: Vacuolization is defined as the presence of more than one vacuole (defined as a clear, round structure in the INL of the retina of at least 30 microns in diameter) compared to baseline in either the left or right eye as evaluated by ocular coherence tomography (OCT).
Time Frame: Up to 12 months
Population: The analysis population consisted of all participants who took at least one dose of study medication, and had a baseline and at least one post-baseline vacuolation assessment.
Measure: Number; unit: participants
Arm/Group | Vorapaxar | Placebo
Number analyzed (Participants) | 91 | 86
participants
  4 months (n=91, n=86) | 1 | 0
  8 months (n=86, n=80) | 1 | 0
  12 months (n=77, n=78) | 0 | 0

2. Secondary Outcome: Number of Participants Who Have a Decrease in Visual Acuity Score of at Least Seven Letters From Baseline
Description: Visual acuity was assessed in both eyes by best corrected visual acuity following standardized refraction. The best corrected visual acuity score is the number of letters on a standard visual acuity testing chart read correctly by a participant. A decrease in best corrected visual acuity score in the left and/or right eye indicates a worsening of vision.
Time Frame: Baseline and 4, 8 and 12 months
Population: The analysis population consisted of all participants who took at least one dose of study medication, and had a baseline and at least one post-baseline visual acuity score.
Measure: Number; unit: participants
Arm/Group | Vorapaxar | Placebo
Number analyzed (Participants) | 90 | 86
participants
  4 months (n=90, n=86) | 10 | 8
  8 months (n=86, n=80) | 10 | 8
  12 months (n=78, n=78) | 7 | 9

3. Secondary Outcome: Number of Participants With Change From Baseline of Center Foveal Thickness of Greater Than 15 Microns as Measured by OCT
Description: Center foveal thickness measured by OCT was evaluated for a change from baseline in greater than 15 microns in either the left or right eye.
Time Frame: Baseline and 4, 8 and 12 months
Population: The analysis population consisted of all participants who took at least one dose of study medication, and had a baseline and at least one post-baseline center point thickness assessment by OCT.
Measure: Number; unit: participants
Arm/Group | Vorapaxar | Placebo
Number analyzed (Participants) | 91 | 86
participants
  4 months (n=91, n=86) | 27 | 28
  8 months (n=86, n=80) | 23 | 26
  12 months (n=77, n=78) | 19 | 29

4. Secondary Outcome: Change From Baseline in the Numerical Score of Graded Abnormalities as Measured by OCT
Description: Individual OCT abnormalities were scored as 0=not present or 1=present. The total number of possible abnormalities present was 84 (42 possible abnormalities per eye). Data are for the left and right eyes combined (score range: 0 to 84). Change from Baseline at a given timepoint was calculated as Timepoint Score minus Baseline Score. A smaller score indicates fewer graded abnormalities.
Time Frame: Baseline and 4, 8 and 12 months
Population: The analysis population consisted of all participants who took at least one dose of study medication, and had a baseline and at least one post-baseline numerical score of graded abnormalities assessment by OCT.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Vorapaxar | Placebo
Number analyzed (Participants) | 92 | 87
score on a scale
  Baseline score (n=92, n=87) | 3.1 (0.3) | 3.4 (0.4)
  4 months change (n=91, n=86) | 0.2 (0.3) | 0.7 (0.3)
  8 months change (n=86, n=80) | 0.6 (0.3) | 0.9 (0.3)
  12 months change (n=77, n=78) | 0.2 (0.3) | 0.0 (0.3)

5. Secondary Outcome: Change From Baseline in the Numerical Score of Graded Abnormalities as Measured by Fundus Photography
Description: Individual fundus photography abnormalities were scored as 0=not present or 1=present. The total number of possible abnormalities present was 48 (24 possible abnomalities per eye). Data are for the left and right eyes combined (score range: 0 to 48). Change from Baseline at a given timepoint was calculated as Timepoint Score minus Baseline Score. A smaller score indicates fewer graded abnormalities.
Time Frame: Baseline and 4, 8 and 12 months
Population: The analysis population consisted of all participants who took at least one dose of study medication, and had a baseline and at least one post-baseline numerical score of graded abnormalities assessment as measured by fundus photogrpahy.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Vorapaxar | Placebo
Number analyzed (Participants) | 91 | 87
score on a scale
  Baseline score (n=91, n=87) | 4.1 (0.4) | 3.9 (0.4)
  4 months change (n=90, n=86) | -0.2 (0.4) | -0.4 (0.3)
  8 months change (n=86, n=80) | -0.4 (0.4) | -0.6 (0.4)
  12 months change (n=76, n=77) | -0.6 (0.5) | -0.3 (0.5)

ADVERSE EVENTS:
Description: Participant safety data collected on the eCRF for this study (SCH 530348 P05183) were limited to ocular test results. These ocular test results were not captured as adverse events, but were captured as part of outcome measures. All other participant adverse events were collected under the Study SCH 530348 P04737 (NCT00526474) parent protocol.
Arm/Group | Vorapaxar | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the study.